CLINICAL TRIAL: NCT03508687
Title: An Investigator-Initiated Open-Label, Randomized Study of Gemcabene in Adults With Familial Partial Lipodystrophy Disease (FPLD)
Brief Title: Study of Gemcabene in Adults With FPLD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elif Oral (Other)
Responsible Party: Sponsor-Investigator, Elif Oral, Professor of Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HUM00130803
Record Dates: First submitted 2018-04-03; First posted 2018-04-26 (Actual); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Familial Partial Lipodystrophy; Hypertriglyceridemia; Fatty Liver; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Lipodystrophy, Familial Partial; Hypertriglyceridemia; Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — gemcabene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: 300 mg Gemcabene daily week 12-24 (Experimental): Patients took Gemcabene 300mg daily for weeks 1-12. After 12 weeks, at visit T4, patients were randomized 1:1 according to pre-generated randomization code. This arm received 300mg Gemcabene daily for 12 weeks total, starting at week 12.
  Interventions: Drug: 300mg Gemcabene
- Group 2: 600mg Gemcabene daily week 12-24 (Experimental): Patients took Gemcabene 300mg daily for weeks 1-12. After 12 weeks, at visit T4, patients were randomized 1:1 according to pre-generated randomization code. This arm received 600mg Gemcabene daily for 12 weeks total, starting at week 12.
  Interventions: Drug: 600mg Gemcabene

INTERVENTIONS:
Drug: 300mg Gemcabene — 300mg Gemcabene
  Arms: Group 1: 300 mg Gemcabene daily week 12-24
Drug: 600mg Gemcabene — 600mg Gemcabene
  Arms: Group 2: 600mg Gemcabene daily week 12-24

SUMMARY:
The overall objective of this study is to assess the efficacy and safety of two dosing regimens of gemcabene (300 mg once daily for 24 weeks or 300 mg daily for 12 weeks followed by 600 mg daily for 12 weeks) in up to eight patients with Familial Partial Lipodystrophy with high triglycerides and Non-Alcoholic Fatty Liver Disease. The study will consist of a six week Wash Out Period, up to a 28 day Screening Period, a 24 week Treatment Period, and a follow-on safety assessment four weeks post final dose. Study participation will last approximately 4 months and includes at least 9 study visits, and can be as many as 11 study visits.

DETAILED DESCRIPTION:
Patients with typical Familial Partial Lipodystrophy Disease (FPLD) have a marked loss of subcutaneous fat from the extremities and trunk accompanied by a variable amount of excess fat deposition in the nonlipodystrophic areas such as the face, chin, back, and intraabdominal regions. Dietary fat restriction and other lifestyle changes are first line therapy to avoid weight gain, critical for effective management of metabolic complications in patients with lipodystrophy. However, despite lifestyle changes and conventional hypoglycemic and hypolipidemic therapies, some FPLD patients continue to have extreme hypertriglyceridemia, hepatic steatosis, and poorly controlled diabetes.Hypertriglyceridemia is a common condition of FPLD and serum triglyceride levels of 250-1999 mg/dL, classified as moderate to severe hypertriglyceridemia, indicate risk for development of very severe hypertriglyceridemia, causative of pancreatitis and hepatic steatosis. In patients such as those with FPLD with severe or very severe hypertriglyceridemia, fibrates, omega-3 fatty acids (OMG-3) and occasionally niacin are first-line therapy. Non-alcoholic fatty liver disease (NAFLD) is often associated with FPLD. The spectrum of NAFLD associated with FPLD which appears to be more frequent than what is seen in common Type 2 diabetes and appears more severe than common forms of NAFLD and very often associated with NASH. The etiology for the latter is not clear, however, the fact that a mouse model of liver specific laminopathy develops NASH in a cell -autonomous manner suggests that the specific cellular defects seen in FPLD may play a role in the development of NAFLD/NASH. Triglyceride content in the liver is regulated by fatty acid uptake as well as fatty acid and VLDL production rates. Derangements in these processes, such as excessive production of fatty acids and triglycerides that can occur with excessive carbohydrate consumption contribute to NAFLD. Patients with NAFLD compared to controls, present with an atherogenic dyslipidemic profile, characterized by increased serum levels of triglycerides, ApoB, VLDL-C, and LDL-C with a proportionally greater content of small dense LDL-C (sdLDL-C) 18-20. NAFLD is also associated with aberrant nuclear receptor function and systemic inflammation. NAFLD can progress to NASH. NASH is marked by hepatocyte ballooning and liver inflammation, which may progress to scarring and irreversible damage. Macro and microscopically, NASH is characterized by lobular and/or portal inflammation, varying degrees of fibrosis, hepatocyte death and pathological angiogenesis. At its most severe, NASH can progress to cirrhosis, hepatocellular carcinoma (HCC) and liver failure. It is estimated that 20-33% NAFLD patients will progress to NASH, with about 5% ultimately progressing to cirrhosis. Cirrhosis has a reported 7- to 10-year mortality of 12-25%. As NAFLD and NASH continue to be a growing epidemic, gemcabene's clinical and preclinical data suggest that this novel agent may provide benefit to patients with the diagnosis of NAFLD and/or NASH. As such, further development of gemcabene may help meet an unmet medical need in these patient populations. In Phase 2 studies, gemcabene has shown triglyceride lowering from 20 to > 50% based on dose and severity of hypertriglyceridemia and lowering in hsCRP of up to 50%. Additionally, in animal and cell based models, gemcabene studies have provided evidence demonstrating: reduction in de-novo lipogenesis, reduction in intrahepatic TG levels, modulation of inflammation and reduction of the NAFLD activity score, particularly related to hepatic ballooning, steatosis, fibrosis, and collagen accumulation. As such gemcabene may have utility in hypertriglyceridemia of FLP and ultimately in the prevention or treatment of NASH in these patients.

ELIGIBILITY:
* Clinical diagnosis of lipodystrophy based on a lack of body fat in a partial fashion assessed by physical examination, and at least 1 MAJOR criterion (below):
* Low skinfold thickness in anterior thigh by caliper measurement: men (≤ 10 mm) and women (≤ 22 mm) OR
* Historic genetic diagnosis of familial partial lipodystrophy (e.g. mutations in LMNA, PPAR-γ, AKT2, or PLIN1 genes) as supported by source documentation
* Hepatic steatosis (>10% - Stage 2 or 3) as demonstrated by MRI-PDFF;
* Alcohol intake of less than 20 g per day in females and 30 g per day in males (one 12 oz beer, one glass of wine, or 2 oz of spirits or liquor equals roughly 10 g of alcohol;
* Mean fasting triglyceride value ≥ 250 mg/dL at the Screening Visit;
* Background lipid lowering medications must be stable for at least 6 weeks prior to the Screening Visit;
* Women patients must not be pregnant or lactating and women of child-bearing potential must agree to use acceptable methods of contraception throughout the duration of the study and for 30 days after the last dose of study drug. Male patients must agree to use contraception by means of a condom and may not donate sperm throughout the duration of the study and for 8 days after the last dose of study drug.
* Weight greater than 50 kg (~110 lbs); with a body mass index (BMI) of no more than 45 kg/m²;
* Have not used a fibrate with in the last 6 weeks and/or thiazolidinediones (TZDs) within the last 12 weeks prior to the Screening visit.
* Do not have a hypersensitivity or a history of significant reactions of fibrates.
* Are not currently taking potent CYP3A4 inhibitors such as itraconazole or a macrolide antibiotic.
* Have a condition or finding which, in the opinion of the Investigator, would compromise the patient's safety or participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Oral, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 300 mg Gemcabene Daily Week 1-24: Patients will take Gemcabene 300mg daily for weeks 1-12. After 12 weeks, at visit T4, patients will be randomized 1:1 according to pre-generated randomization code to either of the following groups. Group 1: Gemcabene 300mg daily for weeks 12-24. Group 2: Gemcabene 600mg daily for weeks 12-24. This arm will receive 300mg Gemcabene daily for 12 weeks total, starting at week 12.
  300mg Gemcabene: 300mg Gemcabene
- Group 2: 600mg Gemcabene Daily Week 12-24: Patients will take Gemcabene 300mg daily for weeks 1-12. After 12 weeks, at visit T4, patients will be randomized 1:1 according to pre-generated randomization code to either of the following groups. Group 1: Gemcabene 300mg daily for weeks 12-24. Group 2: Gemcabene 600mg daily for weeks 12-24. This arm will receive 600mg Gemcabene daily for 12 weeks total, starting at week 12.
  600mg Gemcabene: 600mg Gemcabene
Period: Overall Study
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24 | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 56 [53 to 59] | 52 [38 to 63] | 54 [38 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Fasting Serum Triglycerides [Mean (Full Range); unit: mg/dL] — Patient's fasting serum triglycerides measured in mg/dL.
  mg/dL | 283 [260 to 307] | 790 [255 to 1557] | 587 [255 to 1557]

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Serum Triglyceride (at 12 Weeks)
Description: This is measured by percent change in fasting serum triglyceride from baseline to week 12
Time Frame: Baseline to week 12
Measure: Mean (Full Range); unit: percent change
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
percent change | -0.44 [-41.27 to 40.38] | -20.27 [-53.98 to 12.77]
Statistical Analysis 1: Comparison: Group 1: 300 mg Gemcabene Daily Week 1-24 vs Group 2: 600mg Gemcabene Daily Week 12-24; Test type: Other; p = 0.517, t-test, 2 sided — paired t test; baseline vs. week 12 (n = 5)
Statistical Analysis 2: Comparison: Group 1: 300 mg Gemcabene Daily Week 1-24 vs Group 2: 600mg Gemcabene Daily Week 12-24; Test type: Other; p = 0.345, Wilcoxon (Mann-Whitney); Wilcoxon Signed Ranks Test (n = 5)

2. Secondary Outcome: Change in Fasting Serum Triglycerides (Through 24 Weeks)
Description: This is measured by change in fasting serum triglyceride from baseline to average of weeks 6 and 12, and week 24 and change in fasting serum triglyceride from baseline to week 12
Time Frame: Baseline, week 6 and week 12, week 24
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
mg/dL
  Baseline to average of W6, W12, W24 | 9.25 [-68.50 to 87.00] | -126.22 [-252.17 to -10.50]
  Baseline to W12 | -10.75 [-126.50 to 105.00] | -189.33 [-305.00 to 32.50]

3. Secondary Outcome: Percent Change in Fasting Serum Triglycerides (Through 24 Weeks)
Description: This is measured by percent change in fasting serum triglyceride from baseline to average of weeks 6 and 12, and week 24 and change in fasting serum triglyceride from baseline to week 12
Time Frame: Baseline, week 6 and week 12, week 24
Measure: Mean (Full Range); unit: percent change
Groups:
- Group 1: 300 mg Gemcabene Daily Week 12-24: After 12 weeks, at visit T4, patients will be randomized 1:1 according to pre-generated randomization code to either of the following groups. Group 1: Gemcabene 300mg daily for weeks 12-24. Group 2: Gemcabene 600mg daily for weeks 12-24. This arm will receive 300mg Gemcabene daily for 12 weeks total, starting at week 12.
  300mg Gemcabene: 300mg Gemcabene
- Group 2: 600mg Gemcabene Daily Week 12-24: After 12 weeks, at visit T4, patients will be randomized 1:1 according to pre-generated randomization code to either of the following groups. Group 1: Gemcabene 300mg daily for weeks 12-24. Group 2: Gemcabene 600mg daily for weeks 12-24. This arm will receive 600mg Gemcabene daily for 12 weeks total, starting at week 12.
  600mg Gemcabene: 600mg Gemcabene
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 12-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
percent change
  Baseline to average of W6, W12, and W24 | 5.56 [-22.35 to 33.46] | -18.91 [-45.15 to -4.15]
  Baseline to Week 12 | -0.44 [-41.27 to 40.38] | -19.91 [-52.91 to 12.77]

4. Secondary Outcome: Change in Liver Fat Content as Measured by Magnetic Resonance Imaging - Protein Density Fat Fraction (MRI-PDFF)
Description: This is measured by change in liver fat content using Magnetic Resonance Imaging - Protein Density Fat Fraction (MRI-PDFF) from baseline to week 12 and week 24
Time Frame: Baseline, week 12, week 24
Measure: Mean (Full Range); unit: % PDFF
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
% PDFF
  Baseline to Week 12 | 2.71 [0.37 to 5.05] | 1.01 [-4.22 to 7.76]
  Baseline to Week 24 | 12.75 [9.53 to 15.96] | -1.27 [-8.54 to 8.20]

5. Secondary Outcome: Percent Change in Liver Fat Content as Measured by Magnetic Resonance Imaging - Protein Density Fat Fraction (MRI-PDFF)
Description: This is measured by percent change in liver fat content using Magnetic Resonance Imaging - Protein Density Fat Fraction (MRI-PDFF) from baseline to week 12 and week 24
Time Frame: Baseline, week 12, week 24
Measure: Mean (Full Range); unit: percent change in liver fat
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
percent change in liver fat
  Baseline to Week 12 | 25.66 [2.10 to 49.22] | 11.57 [-31.73 to 69.22]
  Baseline to Week 24 | 104.88 [54.21 to 155.56] | -3.36 [-64.21 to 73.15]

6. Secondary Outcome: Change in Liver Fibrosis
Description: This is measured by change in liver fibrosis using MR-elastography from baseline to week 12 and week 24
Time Frame: Baseline, Week 12, and Week 24
Population: Percentage of change in Preliminary Hepatic Fat-Fraction (PDFF)
Measure: Mean (Full Range); unit: kPA
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
kPA
  Baseline to Week 12 | -0.63 [-0.63 to -0.63] | 0.96 [-0.05 to 1.73]
  Baseline to Week 24 | -0.03 [-0.45 to 0.39] | .45 [0.07 to 2.47]

7. Secondary Outcome: Percent Change in Liver Fibrosis
Description: This is measured by percent change in liver fibrosis using MR-elastography from baseline to week 12 and week 24
Time Frame: Baseline, Week 12, and Week 24
Measure: Mean (Full Range); unit: percent change in fibrosis
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
percent change in fibrosis
  Baseline to Week 12 | -19.07 [-19.87 to -18.26] | 27.84 [-2.04 to 62.10]
  Baseline to Week 24 | -0.37 [-13.04 to 12.30] | 41.55 [2.86 to 88.53]

8. Secondary Outcome: Change in NAS (Non-alcoholic Steatohepatitis)
Description: This is measured by change in NAS via non-alcoholic fatty liver disease activity score. NAS is the unweighted sum of steatosis, lobular inflammation and hepatocyte ballooning from baseline to week 24. Total NAS scores can range from 0 to 8. The higher the NAS score, the more severe the liver disease.
Time Frame: Baseline to week 24
Population: Liver biopsy was performed in two participants at baseline (1 subject in group-1 and another subject in group-2).
  Paired liver biopsy was only available for the subject in group-1.
Measure: Mean (Full Range); unit: scores on a scale (NAFLD activity score)
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 1 | 1
scores on a scale (NAFLD activity score) | 2 [2 to 2] | NA [NA to NA] — Paired liver biopsy was not available for the subject in this group, week 24 data was not collected.

9. Secondary Outcome: Percent Change in NAS (Non-alcoholic Steatohepatitis)
Description: as for outcome 8
Time Frame: Baseline to week 24
Measure: Mean (Full Range); unit: percent change
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 1 | 1
percent change | 100 [100 to 100] | NA [NA to NA] — Paired liver biopsy was not available for the subject in this group. Subject 602-007 (group-2): Baseline NAS = 3, week 24 not available.

10. Secondary Outcome: Change in Cholesterol
Description: This will be measured by change in total, HDL and LDL levels in mg/dL
Time Frame: Baseline, week 6 and week 12, week 24
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
mg/dL
  Total Cholesterol Baseline to Week 12 | -7.00 [-24.00 to 10.00] | -16.67 [-39.00 to 0]
  Total Cholesterol Baseline to Week 24 | 20.50 [13.00 to 28.00] | 23.67 [-19.00 to 82.00]

11. Secondary Outcome: Percent Change in Cholesterol
Description: This will be measured as percent change in total, HDL and LDL levels in mg/dL.
Time Frame: Baseline, week 6 and week 12, week 24
Measure: Mean (Full Range); unit: percent change
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
percent change
  Total Cholesterol Baseline to Week 12 | -4.08 [-14.16 to 6.29] | -7.61 [-19.21 to 0]
  Total Cholesterol Baseline to Week 24 | 12.52 [8.18 to 16.87] | 6.73 [-10.73 to 26.97]

12. Secondary Outcome: Change in Apolipoprotein
Description: This will be measured by change in apolipoprotein A and B in mg/dL
Time Frame: Baseline, week 6 and week 12, week 24
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
mg/dL
  Apolipoprotein B Baseline to Week 12 | -4.35 [-17.02 to 8.33] | -8.76 [-27.00 to 5.29]
  Apolipoprotein B Baseline to Week 24 | 6.74 [-5.73 to 19.22] | 7.57 [-13.89 to 31.47]

13. Secondary Outcome: Percent Change in Apolipoprotein
Description: This will be measured by percent change in apolipoprotein A and B in mg/dL
Time Frame: Baseline, week 6 and week 12, week 24
Population: % Change in participants in group A and group B
Measure: Mean (Full Range); unit: percent change
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
percent change
  Apolipoprotein B Baseline to Week 12 | -5.38 [-21.33 to 10.57] | -6.04 [-19.90 to 4.79]
  Apolipoprotein B Baseline to Week 24 | 8.60 [-7.18 to 24.38] | 5.02 [-10.24 to 20.66]

14. Secondary Outcome: Change in High-Sensitivity C-Reactive Protein (hsCRP)
Description: This is measured by change in high-sensitivity C-reactive protein (hsCRP) from baseline to weeks 12 and week 24
Time Frame: Baseline, week 12, week 24
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
mg/dL
  hsCRP Baseline to Week 12 | -0.70 [-1.30 to -0.10] | -0.33 [-2.40 to 0.80]
  hsCRP Baseline to Week 24 | 0.15 [0.10 to 0.20] | 0.77 [-2.00 to 2.90]

15. Secondary Outcome: Percent Change in High-Sensitivity C-Reactive Protein (hsCRP)
Description: This is measured by percent change in high-sensitivity C-reactive protein (hsCRP) from baseline to weeks 12 and week 24
Time Frame: Baseline, week 12, week 24
Measure: Mean (Full Range); unit: percent change
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
percent change
  hsCRP Baseline to W12 | -42.36 [-72.22 to -12.50] | 3.71 [-63.16 to 57.14]
  hsCRP Baseline to W24 | 15.28 [5.56 to 25.00] | 43.41 [-52.63 to 100.00]

16. Secondary Outcome: Change in Alanine Aminotransferase (ALT)
Description: This is measured by change in alanine aminotransferase (ALT) from baseline to weeks 12 and week 24
Time Frame: Baseline, week 12, week 24
Measure: Mean (Full Range); unit: IU/L
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
IU/L
  ALT Baseline to Week 12 | 2.50 [1.00 to 4.00] | 13.33 [-13.00 to 41.00]
  ALT Baseline to Week 24 | 22.50 [14.00 to 31.00] | 40.67 [-11.00 to 89.00]

17. Secondary Outcome: Percent Change in Alanine Aminotransferase (ALT)
Description: This is measured by percent change in alanine aminotransferase (ALT) from baseline to weeks 12 and week 24
Time Frame: Baseline, week 12, week 24
Measure: Mean (Full Range); unit: percent change
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
percent change
  ALT Baseline to W12 | 6.32 [3.13 to 9.52] | 40.10 [-38.24 to 141.38]
  ALT Baseline to W24 | 58.78 [43.75 to 73.81] | 82.17 [-32.35 to 151.72]

18. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: This is measured by change in aspartate aminotransferase (AST) from baseline to weeks 12 and week 24
Time Frame: Baseline, week 12, week 24
Measure: Mean (Full Range); unit: IU/L
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
IU/L
  AST Baseline to Week 12 | 6.00 [2.00 to 10.00] | 8.00 [-10.00 to 32.00]
  AST Baseline to Week 24 | 11.00 [4.00 to 18.00] | 62.67 [-7.00 to 116.00]

19. Secondary Outcome: Percent Change in Aspartate Aminotransferase (AST)
Description: This is measured by percent change in aspartate aminotransferase (AST) from baseline to weeks 12 and week 24
Time Frame: Baseline, week 12, week 24
Measure: Mean (Full Range); unit: percent change
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
Number analyzed (Participants) | 2 | 3
percent change
  AST Baseline to W12 | 19.25 [9.09 to 29.41] | 25.44 [-33.33 to 106.67]
  AST Baseline to W24 | 35.56 [18.18 to 52.94] | 160.41 [-23.33 to 386.67]

ADVERSE EVENTS:
Time Frame: 28 weeks (24 week Treatment Period, and a follow-on safety assessment 4 weeks post final dose)
Arm/Group | Group 1: 300 mg Gemcabene Daily Week 1-24 | Group 2: 600mg Gemcabene Daily Week 12-24
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 300 mg Gemcabene Daily Week 1-24 (N=2) | Group 2: 600mg Gemcabene Daily Week 12-24 (N=3)
Vertigo (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 300 mg Gemcabene Daily Week 1-24 (N=2) | Group 2: 600mg Gemcabene Daily Week 12-24 (N=3)
Increase in liver fat (Hepatobiliary disorders) | 2 (2) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 1 (1)
Increased Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis of thumb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitis on R finger (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Increase in Creatinine Phosphokinase (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Increased Hunger (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Increased Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 1 (1)
Pain from Liver Bx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sore Throat (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Body Pain (General disorders) | 0 (0) | 1 (1)
Decreased EGFR non-black (Renal and urinary disorders) | 0 (0) | 1 (1)
dizzyness 'spell' has history of these last episode ago 1 year (Nervous system disorders) | 0 (0) | 1 (1)
Dry skin itchniness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fall down steps (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (migraine) (Nervous system disorders) | 0 (0) | 1 (1)
HSV Outbreak (Infections and infestations) | 0 (0) | 1 (1)
hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
increase in calcium level (lab) (Endocrine disorders) | 0 (0) | 1 (1)
Increase in fatigue (General disorders) | 0 (0) | 1 (1)
Increased Blood Sugars (Endocrine disorders) | 0 (0) | 1 (1)
Increased Creatinine (Renal and urinary disorders) | 0 (0) | 2 (2)
increased CRP (Immune system disorders) | 0 (0) | 1 (1)
Increased diabetic neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Increased GGTP (Hepatobiliary disorders) | 0 (0) | 2 (2)
Increased headaches (Nervous system disorders) | 0 (0) | 1 (1)
increased liver enzymes (Hepatobiliary disorders) | 0 (0) | 2 (3)
increased pain hips (arthritis) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Increased stress levels (General disorders) | 0 (0) | 1 (1)
Lesion L side of mouth (Investigations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Pain increased knees both (arthritis bath) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder soreness/stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
upper right quadrant pain of abdomen (General disorders) | 0 (0) | 1 (1)
vomited (intermittent) (Gastrointestinal disorders) | 0 (0) | 1 (1)
weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The expected number of study subjects (8), was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT03508687/Prot_SAP_000.pdf